CLINICAL TRIAL: NCT05092763
Title: A Pilot Study of Prehabilitation During the Neoadjuvant Window of Opportunity in Older Women With Ovarian Cancer (FIT4SURGERY)
Brief Title: Prehabilitation During the Neoadjuvant Window of Opportunity in Older Women With Ovarian Cancer
Acronym: FIT4SURGERY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Emma Barber, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00215518
Record Dates: First submitted 2021-08-13; First posted 2021-10-26 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Cancer; Neoadjuvant Chemotherapy; Prehabilitation
Keywords: ovarian cancer; neoadjuvant chemotherapy; chemotherapy; physical activity; prehabilitation
MeSH Terms: conditions — Ovarian Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FIT4SURGERY Intervention (Experimental): The Fit4Surgery intervention consists of the FitBit Inspire HR device, the Fit4Surgery mobile app, and weekly coaching calls.
  Interventions: Behavioral: FIT4SURGERY
- Healthy Lifestyle Control (Active Comparator): The Healthy Lifestyle Control group engages in their usual activities and receives education about physical activity and a healthy lifestyle for ovarian cancer patients. They receive weekly check in calls.
  Interventions: Behavioral: Healthy Lifestyle Control

INTERVENTIONS:
Behavioral: FIT4SURGERY — The Fit4Surgery intervention consists of the FitBit Inspire HR device, the Fit4Surgery mobile app, and weekly coaching calls. Patients are asked to wear the Fitbit through the entire 9-12 weeks in which they are receiving neoadjuvant chemotherapy both when asleep and when awake. Patients are taught how to understand the Fitbit outputs on the application, for example, understanding how to monitor their steps and heart rate. Caregivers are also be encouraged to assist patients. Patients are provided with information about the benefits of physical activity and effective behavior change strategies for incorporating physical activity into their daily lives. These include things such as short bouts of activity by walking around the room during commercial breaks or planning to be dropped off a short walk from a destination.
  Arms: FIT4SURGERY Intervention
Behavioral: Healthy Lifestyle Control — Participants assigned to this study arm are instructed to go about their usual activities and receive education about physical activity and a healthy lifestyle for ovarian cancer patients. They are encouraged to download the free Cancer.Net mobile app and visit the cancer.net website for educational materials related to ovarian cancer and survivorship. At the end of the 9-12 week intervention, participants in the Healthy Lifestyle group receive a Fitbit for their optional, personal use after surgery.
  Arms: Healthy Lifestyle Control

SUMMARY:
The purpose of this study is to test the effectiveness of a home-based, patient-tailored intervention, FIT4SURGERY, to promote physical activity among women with ovarian cancer undergoing neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Ovarian cancer is the deadliest gynecologic cancer with 5-year survival rates of approximately 48%. Standard of care treatment is grueling, requiring a radical "debulking" surgery and 5 months of chemotherapy. Cytoreductive surgery for ovarian cancer is often extensive, due to the necessary removal of all visible cancer. This radical surgery results in major postoperative complication rates as high as 50% in prospective clinical trials, and 75% occur within 2 weeks of surgery. Half of women are greater than 60 years-old and have high rates of hospital readmission and postoperative complications. Aside from immediate morbidity and mortality related to surgery itself, postoperative complications, such as anastomotic leak, sepsis, or pelvic abscess, can delay the onset of adjuvant chemotherapy, resulting in decreased survival. These postoperative complications also lead to increased discharge to a non-home setting, decreased quality of life, increased costs, and mortality.

Although all patients with ovarian cancer undergo this treatment schedule, older women are at particularly high risk for adverse events. Among women with ovarian cancer, more than 50% are over the age of 60 and up to 40% of these older women are defined as frail. Both age and frailty have been shown to be independent predictors of surgical complications, chemotherapy complications, as well as under-treatment with chemotherapy, resulting in inferior cancer-specific survival. Additionally, the definition of aging contains mechanisms beyond the chronological age of the patient. Both a cancer diagnosis and receipt of chemotherapy lead to synergistic biologic and physiologic changes that accelerate aging and increase frailty. Many older women with ovarian cancer are treated with neoadjuvant chemotherapy which is delivered in 3-4 cycles prior to surgery and this time period provides an optimal window to intervene to improve high-risk older patients' surgical outcomes.

Prehabilitation is the process of enhancing an individual's functional capacity prior to a forthcoming stressor, such as a major surgery, with the goal of improving postoperative outcomes. Prehabilitation programs are multimodal and can involve medical optimization, preoperative physical exercise, nutritional support and stress/anxiety reduction. Benefits of prehabilitation include reduced length of stay, fewer postoperative complications and improved postoperative pain. Even small increases in light physical activity or reducing sedentary time has been shown to slow or halt functional decline and improve quality of life. Among advanced cancer patients, physical activity interventions have been shown to be safe and feasible. They have also been associated with improved aerobic capacity, increased strength, and increased physical function. These parameters are important in older ovarian cancer patients to prevent functional decline, reduce frailty, and decrease surgical morbidity.

However, not all prehabilitation interventions or physical activity interventions are effective. There are populations that do not have sufficient time prior to surgery to have a meaningful change in activity or nutrition, this is especially true for cancer patients who often have a short window between diagnosis and surgery. Furthermore, many physical activity interventions in the pre-operative period have used structured, in-person, professionally-led programs with high intensity activity that may not be appropriate for the changing symptom burden of older ovarian cancer patients undergoing chemotherapy.

Instead of a one-size fits all approach, the American Cancer Society recommends that patients with advanced cancer engage in physical activity tailored to their capability. A recent systematic review and meta-analysis of prehabilitation in cancer patients undergoing abdominal operations noted that data specific to older patients are sparse. This study seeks to address this critical research gap by testing a home-based, patient-tailored, physical activity prehabilitation program (FIT4SURGERY) among older women with ovarian cancer undergoing neoadjuvant chemotherapy.

Physical activity has been shown to improve functional health and energy balance as well as decrease rates of frailty and sarcopenia, important prognostic factors prior to surgery, especially for older adults, and important prognostic factors for ovarian cancer. Increasing physical activity and motivating behavior change is difficult and many preoperative physical activity interventions have not utilized techniques and frameworks which have been successfully used among patients with chronic diseases. Social cognitive theory (SCT) is a framework which has been successfully used to design physical activity inventions that lead to behavior change. SCT has three main components, self-monitoring, self-judgment and self-evaluation which all contribute to self-regulation which is ultimately what drives behavior change. Behavioral interventions using SCT frameworks have been studied in healthy participants including cancer survivors, and have been shown to increase physical activity. Among women with metastatic breast cancer undergoing chemotherapy, an mHealth behavioral physical activity intervention consisting of a wearable activity tracker to provide direct feedback and a mobile app with motivational messaging, has been implemented by our research group. This study examines a modified version of this intervention, as prehabilitation, for the older ovarian cancer patient, as SCT-driven physical activity interventions have not been studied in a preoperative population.

Compared to the gold standard of professionally led, physical activity interventions, interventions via phone and email have been shown to be potentially as effective as more resource intensive interventions at increasing physical activity. Interventions using mHealth app-based platforms have also been shown to increase physical activity. Specifically, for older patients with ovarian cancer undergoing chemotherapy, interventions using wearable devices may be useful because they are home-based, easy to use, give immediate feedback, and use technology most patients already own. Caregivers can also be enlisted to help patients; activating social support for physical activity. Wearable devices allow for remote monitoring of participants and prevent the need for in-person visits which may be difficult for patients undergoing chemotherapy particularly during the COVID-19 pandemic. Furthermore, Fit4Surgery incorporates daily reported symptom burden into activity goals as symptoms can wax and wane during treatment. Such a tailored, home-based, patient-specific approach that facilitates the gradual and safe adoption of physical activity that can be supported by caregivers is ideal for older ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Female; ≥ 60 years of age
* Diagnosed with ovarian, fallopian tube or primary peritoneal cancer and undergoing planned neoadjuvant chemotherapy and are expecting to undergo planned surgery
* Fluent in spoken and written English
* Own a smartphone
* Have access to the internet to complete assessments

Exclusion Criteria:

* Patients receiving planned chemotherapy only
* Patients with uncontrolled cardiovascular disease, who are non-ambulatory, or who have severe cognitive or functional limitations precluding their ability to participate in a physical activity intervention
* Pregnant women or prisoners
* Patients whose oncologist has not provided clearance for their participation

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are evaluable for both baseline and post-intervention assessments | Through study completion, average of 9-12 weeks
  Evaluability will be measured for all patients enrolled in the study regardless of intervention assignment. Patients will be considered evaluable if they complete both the pre-intervention baseline assessments (frailty, PROs) and the post-intervention pre-surgery assessments. The proportion of patients evaluable, according to the above definition, over all patients enrolled will be calculated.
Proportion of patients who are adherent to the Fit4Surgery intervention measured among those in the Fit4Surgery arm. | Through study completion, average of 9-12 weeks
  Adherence will be measured in the Fit4Surgery arm. Patients will be considered adherent to the Fit4Surgery intervention if they wear their Fitbit for >70% of the days during the study period (i.e., ~44/63 days) and if they meet their physical activity goals (step count) on >70% of the days during the study period. The proportion of patients in the Fit4Surgery arm who are adherent to the intervention, according to the above definition, will be calculated.

SECONDARY OUTCOMES:
Change in frailty | Baseline and once at 9-12 weeks
  Frailty will be assessed at baseline and prior to surgery using the "Fried's phenotype method" in patients in both groups. According to this scale, patients will be categorized as non-frail, pre-frail or frail.
Change in anxiety | Baseline and once at 9-12 weeks
  Anxiety will be measured using "PROMIS anxiety short form 7a" measure.
Change in physical function | Baseline and once at 9-12 weeks
  Physical function will be measured using "PROMIS physical function short form 10a" measure.
Change in fatigue | Baseline and once at 9-12 weeks
  Fatigue will be measured using "PROMIS fatigue short form 7a" measure.
Adverse Events | Once at 9-12 weeks
  The number of adverse events will be recorded and graded according to CTCAE v5.0.
Surgical Complications | 90 days post surgery
  Medical record review will be performed to examine postoperative complications which will be graded using the Clavien-Dindo scale.
Progression free survival | three years post surgery
  Medical records will be reviewed for up to three years to monitor for cancer recurrence.
Overall survival | three years post surgery
  Medical records will be reviewed for up to three years to monitor for overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Barber, MD, MS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No